CLINICAL TRIAL: NCT00648141
Title: A 12-Week Symptomatic Effect Evaluation to Compare Celecoxib 200 mg QD, Celecoxib 200 mg BID and Diclofenac 75 mg SR BID in Patients With Ankylosing Spondylitis
Brief Title: Safety and Efficacy of Celecoxib Versus Diclofenac in the Treatment of Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COXA-0508-243; A3191098
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-03

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Celecoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: Celecoxib
- B (Experimental)
  Interventions: Drug: Celecoxib
- C (Active Comparator)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Celecoxib — 200 mg oral capsule once daily for 12 weeks
  Arms: A
Drug: Celecoxib — 200 mg oral capsule twice daily for 12 weeks
  Arms: B
Drug: Diclofenac — 75 mg oral capsule twice daily for 12 weeks
  Arms: C

SUMMARY:
To compare the safety and efficacy of once-daily and twice-daily celecoxib versus diclofenac for the treatment of ankylosing spondylitis

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis defined according to modified New York criteria, and with axial involvement
* Requiring daily treatment with nonsteroidal anti-inflammatory drugs during the previous 30 days

Exclusion Criteria:

* Patients with inflammatory enterophathy, and with extra-articular manifestations
* Patients with known vertebral compression
* Received corticosteroids 6 weeks prior to the baseline visit; patients on stable dose of prednisolone equivalents ≤ 10 mg/ day for at least 14 days before randomization were permitted

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2003-01; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in global pain intensity as assessed by visual analog scale (VAS) | Week 12
Responder rates, defined as 50% improvement in VAS from baseline | Week 12

SECONDARY OUTCOMES:
Patient's and physician's global assessment of disease activity | Weeks 1, 2, 6, and 12
Spinal pain | Weeks 1, 2, 6, and 12
Short Form-12 | Weeks 1, 2, 6, and 12
Adverse events | Week 12
Physical evaluation | Week 12
Laboratory tests | Week 12
Nocturnal pain | Weeks 1, 2, 6, and 12
Composite Bath Ankylosing Spondylitis Disease Activity Index | Weeks 1, 2, 6, and 12
Bath Ankylosing Spondylitis Metrology Index | Weeks 1, 2, 6, and 12
Change from baseline in C-reactive protein measurement | Week 12
Responder rates, defined as 50% improvement in VAS from baseline | Weeks 1, 2, and 6
Mobility parameters | Weeks 1, 2, 6, and 12
Change from baseline in Assessments in Ankylosing Spondylitis 20 score | Weeks 1, 2, 6, and 12
Change from baseline in global pain intensity | Weeks 1, 2, and 6
Bath Ankylosing Spondylitis Functional Index | Weeks 1, 2, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- Germany (41):
  - Pfizer Investigational Site, Aachen
  - Pfizer Investigational Site, Bad Aibling
  - Pfizer Investigational Site, Bad Iburg
  - Pfizer Investigational Site, Bad Münder am Deister
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Celle / OT Klein Hehlen
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Darmstadt
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Elmshorn
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Hildesheim
  - Pfizer Investigational Site, Hofheim
  - Pfizer Investigational Site, Hoyerswerda
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Leverkusen
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Neubrandenburg
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Osnabrück
  - Pfizer Investigational Site, Pirna
  - Pfizer Investigational Site, Ratingen
  - Pfizer Investigational Site, Regensburg
  - Pfizer Investigational Site, Remscheid
  - Pfizer Investigational Site, Rheine
  - Pfizer Investigational Site, Rostock
  - Pfizer Investigational Site, Saarbrücken
  - Pfizer Investigational Site, Seesen
  - Pfizer Investigational Site, Surwold
  - Pfizer Investigational Site, Tübingen
  - Pfizer Investigational Site, Villingen-Schwenningen
  - Pfizer Investigational Site, Weener
  - Pfizer Investigational Site, Winsen

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=COXA-0508-243&StudyName=Safety%20and%20Efficacy%20of%20Celecoxib%20Versus%20Diclofenac%20in%20the%20Treatment%20of%20Ankylosing%20Spondylitis